CLINICAL TRIAL: NCT07142954
Title: A Longitudinal, Prospective Epidemiology Study in Alzheimer's Disease: Assessing Neurocognitive and Biomarker Changes and Health Outcomes in Individuals at Risk for Symptoms of Alzheimer's Disease (ANCHOR-AD)
Brief Title: Epidemiology and Biomarker Study in Alzheimer's Disease
Acronym: ANCHOR-AD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 27588; I5T-MC-AACU (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
Keywords: Preclinical Alzheimer's Disease; Primary Prevention
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elevated Plasma P-tau217 Levels (Other): Participants with known elevated plasma P-tau217 levels who are cognitively unimpaired at baseline per self-report.
  Interventions: Other: P-tau217 Test
- Not-Elevated P-tau217 Levels (Other): Participants with known not-elevated plasma P-tau217 levels who are cognitively unimpaired at baseline per self-report.
  Interventions: Other: P-tau217 Test

INTERVENTIONS:
Other: P-tau217 Test — A plasma test measuring phosphorylated tau at Position 217 (P-tau217).

SUMMARY:
Study AACU determines rates of cognitive worsening in participants within elevated and not elevated plasma P-tau217 cohorts.

Participation in AACU will last approximately 7 years.

DETAILED DESCRIPTION:
Study AACU is a non-drug interventional study. The intervention is annual plasma P-tau217 testing. Enrollment is anticipated to be approximately 3400 participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant must self-report unimpaired cognition.
* The participant must have adequate literacy, vision, and hearing for neuropsychological assessments at the time of screening.

Exclusion Criteria:

* Have seen a doctor about memory concerns.
* Have a history or diagnosis of cognitive impairment, or significant other neurodegenerative disease that can affect cognition.
* Are currently enrolled or have previously participated in any Alzheimer's Disease (AD)-related study involving an investigational drug intervention.
* Are currently using or have previously used prescription medications for treatment of mild cognitive impairment (MCI) or dementia such as amyloid targeting therapy (that is, lecanemab, donanemab, aducanumab), cholinesterase inhibitors (for example, benzgalantamine, donepezil, galantamine, rivastigmine), and memantine.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2033-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Time to Cognitive Worsening Within Cohorts as Measured by Cognitive Composite or Any of the Individual Composite Components | Baseline up to 7 years
  Cognitive composite may consist of International Daily Symbol Substitution Test-Medicines (iDSSTm ), International Shopping List Test (ISLT), Continuous Paired Associate Learning Test (CPAL).
  Time to cognitive worsening is defined as a change in cognitive composite score or any of the individual composite components, from baseline at 2 consecutive visits.

SECONDARY OUTCOMES:
Time to Cognitive Worsening Between Groups (Participants Within Elevated and Not-Elevated Plasma P-Tau217) as Measured by Cognitive Composite or Any of the Individual Composite Components | Baseline up to 7 years
  Cognitive composite may consist of iDSSTm, ISLT, and CPAL Time to cognitive worsening is defined as a change in cognitive composite score or any of the individual composite components, from baseline at 2 consecutive visits.
Time to Cognitive Worsening within Cohorts as Measured by Cognitive Function Index (CFI) | Baseline up to 7 years
Time to Cognitive Worsening within Cohorts as Measured by Montreal Cognitive Assessment XpressO version (XpressO) | Baseline up to 7 years
Time to Cognitive Worsening Between Groups as Measured by CFI | Baseline up to 7 years
Time to Cognitive Worsening Between Groups as Measured by XpressO | Baseline up to 7 years
Change from Baseline Within Not-Elevated and Elevated P-tau217 Groups as Measured by Cognitive Composite Score | Baseline, Year 7
Change from Baseline Within Not-Elevated and Elevated P-tau217 Groups as Measured by ISLT | Baseline, Year 7
Change from Baseline Within Not-Elevated and Elevated P-tau217 Groups as Measured by iDSSTm | Baseline, Year 7
Change from Baseline Between Not-Elevated and Elevated P-tau217 Groups as Measured by Cognitive Composite Score | Baseline, Year 7
Change from Baseline Between Not-Elevated and Elevated P-tau217 Groups as Measured by ISLT | Baseline, Year 7
Change from Baseline Between Not-Elevated and Elevated P-tau217 Groups as Measured by iDSSTm | Baseline, Year 7
Weighted Proportion of Participants with Elevated Plasma P-tau217 Levels in US and Japan with Unimpaired Cognition at Baseline | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Care Access - Houston, Houston, Texas, United States
- Japan (2):
  - The University of Tokyo Hospital, Bunkyō City
  - Souseikai Sumida Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No